CLINICAL TRIAL: NCT04462523
Title: Open-label, Single -Center, Prospective Study on the Efficacy and Safety of Intracanalicular Dexamethasone Insert 0.4mg (Dextenza) in the Treatment of Postoperative Pain and Inflammation Following Vitreo-retinal Surgery - The ADHERE Study
Brief Title: DEXTENZA for the Treatment of Postoperative Pain and Inflammation Following Vitreo-retinal Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Patrick R. Oellers, MD (Network)
Collaborators: Ocular Therapeutix, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Patrick R. Oellers, MD, Principal Investigator, Retina Vitreous Surgeons of Central New York, PC
Organization: Retina Vitreous Surgeons of Central New York, PC (Network)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: The ADHERE Study
Record Dates: First submitted 2020-06-24; First posted 2020-07-08 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Vitreo-Retinal Surgery
MeSH Terms: interventions — Calcium Dobesilate; Prednisolone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Masked Sub-investigators to exam subjects at each visit after clinical evaluation for cell and/or flare.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1 Pre-surgery Dextenza insert (Experimental): Ten patients will receive the dexamethasone intracanalicular insert pre-operatively (1 week to 1 days prior to vitreo-retinal surgery). All patients no matter what cohort will receive Gentamicin, antibiotic ophthalmic drops.
  Interventions: Drug: Dextenza 0.4Mg Ophthalmic Insert
- Group 2 Surgery Day Dextenza insert (Experimental): Ten patients will receive dexamethasone intracanalicular insert on the day of surgery. All patients no matter what cohort will receive Gentamicin, antibiotic ophthalmic drops.
  Interventions: Drug: Dextenza 0.4Mg Ophthalmic Insert
- Group 3 Post op Day 1 Dextenza insert (Experimental): Ten patients will receive DEXTENZA insert Day 1 post-operatively. All patients no matter what cohort will receive Gentamicin, antibiotic ophthalmic drops
  Interventions: Drug: Dextenza 0.4Mg Ophthalmic Insert
- Group 4 Topical steroid (Active Comparator): Ten patients will be prescribed standard of care ophthalmic drops, Prednisolone Acetate, and no dexamethasone insert (control group). All patients no matter what cohort will receive Gentamicin, antibiotic ophthalmic drops.
  Interventions: Drug: Topical Prednisolone

INTERVENTIONS:
Drug: Dextenza 0.4Mg Ophthalmic Insert — The insert, containing 0.4 mg of active pharmaceutical product, is placed within the canaliculus to provide a sustained and tapered delivery of drug to the ocular surface over 30 days after a one-time insertion. The attributes of the insert reduce the risks for improper corticosteroid tapering and unwanted peaks and troughs in drug concentration.
  Arms: Group 1 Pre-surgery Dextenza insert; Group 2 Surgery Day Dextenza insert; Group 3 Post op Day 1 Dextenza insert
Drug: Topical Prednisolone — Standard of care topical drop treatment
  Arms: Group 4 Topical steroid

SUMMARY:
The purpose of this study is to evaluate efficacy and safety of Dextenza for the treatment of postoperative pain and inflammation following vitreo-retinal surgery

DETAILED DESCRIPTION:
This prospective, single-center, open-label, investigator-sponsored clinical study seeks to investigate the outcomes of patients undergoing vitro-retinal surgery with the treatment of a dexamethasone intracanalicular insert. All patients in the treatment groups will receive a dexamethasone intracanalicular insert. There will be three experimental groups of patients, varying that time of insertion. Ten patients will receive the dexamethasone intracanalicular insert pre-operatively (1 week to 1 days prior to vitreo-retinal surgery). Ten patients will receive dexamethasone intracanalicular insert on the day of surgery. Ten patients will receive DEXTENZA insert Day 1 post-operatively. Ten patients will be prescribed standard of care ophthalmic drops, Prednisolone Acetate, and no dexamethasone insert (control group). All patients no matter what cohort will receive Gentamicin, antibiotic ophthalmic drops.

ELIGIBILITY:
Inclusion Criteria:

* Any adult patient age 18-99 years who is planned to undergo vitreo-retinal surgery (pars plana vitrectomy with or without scleral buckle).
* If both eyes are involved, both eyes would be eligible for the study.
* Willing and able to comply with clinic visits and study related procedures.
* Willing and able to sign the informed consent form.

Exclusion Criteria:

* Patients under age 18.
* Patients who are pregnant (must be ruled out in women of child-bearing age with pregnancy test).
* Active infectious ocular or systemic disease.
* Patients with active infectious ocular or extraocular disease.
* Patients actively treated with local or systemic immunosuppression
* Use of the following anti-inflammatory or immunomodulating agents (e.g., cyclosporine) systemically, or in the study eye, for the duration of the study (excluding inhalants). Washout periods for medications prior to surgery are as follows:
* Systemic corticosteroids - 2 weeks (see exception 5c)
* Systemic NSAID over 375 mg per day - 2 weeks
* Periocular/intraocular injection of any corticosteroid solution - 4 weeks (see exception 5b)
* Corticosteroid depot/implant in the study eye - 2 months
* Topical ocular corticosteroid - 7 days
* Topical ocular NSAID - 7 days
* Intraoperatively used intraocular steroid (i.e. intravitreal triamcinolone, that is used to transiently highlight the vitreous and removed during vitrectomy) is permissible in study eye.
* Intraoperatively or perioperatively used systemic steroid for the purpose of general anesthesia (as administered by the treating anesthesiologist) is permissible.
* Patients with systemic illness involving abnormalities of the hypothalamic-pituitary-adrenal axis; patients with primary adrenocortical insufficiency or adrenocortical hyperfunction.
* Patients with known hypersensitivity to Dexamethasone.
* Patients with uncontrolled glaucoma.
* Patients with severe disease that warrants critical attention, deemed unsafe for the study by the investigator.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-01-03 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Mean cells as assessed by investigator in anterior chamber of the study eye | Assessed at Day 14
  As measure by Standardization of Uveitis Nomenclature (SUN Scale) (Grade 0 to Grade 4+)
Mean pain as reported by subject in the study eye: Visual Analog Scale | Assessed at Day 28
  As measured by Visual Analog Scale for Pain (VAS Pain) (0% to 100% Scale)

SECONDARY OUTCOMES:
Mean anterior chamber flare | Assessed at Screening, Day 1, Day 4, Day 14, Day 28 and Day 56
  As measure by Standardization of Uveitis Nomenclature (SUN Scale) (Grade 0 to Grade 4+)
Time to absence of cells | Assessed at Screening, Day 1, Day 4, Day 14, Day 28 and Day 56
  As measure by Standardization of Uveitis Nomenclature (SUN Scale) (Grade 0 to Grade 4+)
Time to absence of pain | Assessed at Screening, Day 1, Day 4, Day 14, Day 28 and Day 56
  As measure by Visual Analog Scale for Pain (VAS Pain) (0% to 100% Scale)
Proportion of rescue treatment | Assessed at Screening, Day 1, Day 4, Day 14, Day 28 and Day 56
  As measure by Concomitant Medications as rescue therapy
Assessment of Dextenza ease of insertion | Assessed at Day 1
  As measured by Ease of Use Survey (0=very easy to 10=very hard)

CONTACTS AND LOCATIONS:
Locations (1):
- Retina Vitreous Surgeons of Central New York, PC, Liverpool, New York, United States

REFERENCES:
- [Derived] Ueberroth JA, Oellers PR, Brown J, Rosenberg KI, Breazzano MP. Intracanalicular Dexamethasome Insert after Retinal Surgery: the ADHERE Trial. Ophthalmol Retina. 2023 Sep;7(9):831-833. doi: 10.1016/j.oret.2023.06.011. Epub 2023 Jun 24. No abstract available. PMID 37356492